CLINICAL TRIAL: NCT02909946
Title: Pathway From Functional Disability to Antimicrobial Resistance in Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lona Mody, Principal Investigator, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01AG041780 (NIH)
Record Dates: First submitted 2016-08-16; First posted 2016-09-21 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Multi-antibiotic Resistance
Keywords: multidrug-resistant organisms; nursing home; post-acute care; long-term care; infection control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Active Comparator): NHs randomized to the Intervention Arm will implement a new multi-modal infection control program.
  Interventions: Behavioral: Multi-modal Infection Control Program
- Control Arm (No Intervention): NHs randomized to the Control Arm will continue their current standard infection control practices.

INTERVENTIONS:
Behavioral: Multi-modal Infection Control Program — 1. Standard precautions and hand hygiene for care of all residents. Enhanced barrier precautions including hand hygiene, glove use, and gown use for HCW when providing ADL assistance for residents at highest-risk (caregiver intervention).
  2. Hand hygiene education to residents and families (resident-level intervention).
  3. Standardized bathing practices including using chlorhexidine-based cloths to reduce resident MDRO colonization (resident-level intervention).
  4. Standardized environmental protocol and education to reduce contamination on inanimate objects and surfaces (environmental intervention).
  5. Feedback monthly of facility-level microbial data and new MDRO acquisition rates to infection control practitioners, HCWs, and facility leadership (facility intervention).
  Arms: Intervention Arm

SUMMARY:
Multidrug-resistant organisms (MDROs) are endemic in nursing homes (NHs) with prevalence rates surpassing those in hospitals. The aim of the study is to design and evaluate the effectiveness of a multi-component intervention to reduce new acquisition of MDROs in NH residents. The intervention will incorporate resident-level, environmental, and caregiver based strategies. Using a cluster-randomized study design, three NHs will be randomized to the intervention group and three to the control group. Control NHs will be allowed to continue standard infection prevention practices. Nursing homes will serve as the unit of allocation. Analyses will be performed both at the resident and the cluster level. The primary outcomes of the study are reduction in MDRO prevalence, and reduction in new MDRO acquisition .

DETAILED DESCRIPTION:
The NH intervention will incorporate resident-level, environmental, and caregiver based strategies, including: a. Standard precautions and hand hygiene for care of all residents. Enhanced barrier precautions including hand hygiene, glove use, and gown use for healthcare workers (HCW) when providing activities of daily living (ADL) assistance for residents at highest-risk (caregiver intervention); b. Hand hygiene education to residents and families (resident-level intervention); c. Standardized bathing practices including using chlorhexidine-based cloths to reduce resident MDRO colonization (resident-level intervention); d. Standardized environmental protocol and education to reduce contamination on inanimate objects and surfaces (environmental intervention); e. Feedback monthly of facility-level microbial data and new MDRO acquisition rates to infection preventionists, front-line healthcare personnel, and facility leadership (facility intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Residing in a participating NH facility
* Provided informed consent for participation

Exclusion Criteria:

* Receiving end-of-life care
* Non-English language speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Prevalence density of multidrug-resistant organisms (MDRO) | From enrollment up to 6 months of study followup, or until study withdrawal (discharged from facility, at resident request, death)
  Total number of MDROs isolated across all MDROs and all anatomic sites for all enrolled residents over the duration of the study period

SECONDARY OUTCOMES:
Incidence of multidrug-resistant organisms (MDRO) | From enrollment up to 6 months of study followup, or until study withdrawal (discharged from facility, at resident request, death)
  Total number of MDROs newly acquired (resident not colonized at baseline) isolated across all MDROs for all enrolled residents over the duration of the study period
Incidence of healthcare-associated infections | From enrollment up to 6 months of study followup, or until study withdrawal (discharged from facility, at resident request, death)
  Total number of new infections acquired at the nursing home for all enrolled residents over the duration of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Lona Mody, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan and partner nursing homes, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Wang J, Foxman B, Rao K, Cassone M, Gibson K, Mody L, Snitkin ES. Association of patient clinical and gut microbiota features with vancomycin-resistant enterococci environmental contamination in nursing homes: a retrospective observational study. Lancet Healthy Longev. 2023 Nov;4(11):e600-e607. doi: 10.1016/S2666-7568(23)00188-5. PMID 37924841
- [Derived] Mody L, Gontjes KJ, Cassone M, Gibson KE, Lansing BJ, Mantey J, Kabeto M, Galecki A, Min L. Effectiveness of a Multicomponent Intervention to Reduce Multidrug-Resistant Organisms in Nursing Homes: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2116555. doi: 10.1001/jamanetworkopen.2021.16555. PMID 34269807